CLINICAL TRIAL: NCT01629147
Title: Treatment of Chronic Constipation in Children With Lactobacillus Reuteri (Biogaia): A Prospective Placebo-controlled Trial
Brief Title: Treatment of Chronic Constipation in Children With Lactobacillus Reuteri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Batia Weiss, Director, Division of Pediatric Gastroenterology and Nutrition, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-11-8960-BW-CTIL
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Constipation
Keywords: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biogaia (Experimental): 5 drops containing Lactobacillus reuteri Protectis
  Interventions: Dietary Supplement: Biogaia
- Placebo (Placebo Comparator): - 5 drops identical in appearance and taste
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Biogaia — 5 drops containing Lactobacillus reuteri Protectis
  Arms: Biogaia
Other: Placebo — 5 drops
  Arms: Placebo

SUMMARY:
Lactobacillus reuteri (Biogaia) may be beneficial for treatment of chronic constipation in children 4-10 years of age.

DETAILED DESCRIPTION:
Functional chronic constipation is very common in childhood and is responsible for 20% of the clinic visits in pediatric gastroenterology. Constipation is defined by the Rome III criteria. The symptoms are difficult to treat in part of the patients and cause frustration to the patient and family.

Probiotics are increasingly used in the treatment of functional gastrointestinal disorders, including chronic constipation in adults and children. A recent study revealed that the administration of Lactobacillus reuteri had a positive effect on bowel frequency in infants with chronic constipation.

The study goal is to evaluate Lactobacillus reuteri (Biogaia) for treatment of chronic constipation in children 4-10 years of age, and to examine the influence of Lactobacillus reuteri (Biogaia) on constipation in different age groups of school aged children between 4-10 yrs of age.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 4-10 years old with no underlying chronic illnesses or anatomical abnormalities of the GI tract, with parents agreeing to participate in the study and signing an informed consent.
2. Chronic constipation defined by the Rome III criteria (Must include 2 or more of the following in a child with a developmental age of at least 4 years with insufficient criteria for diagnosis of IBS: 1. Two or fewer defecations in the toilet per week. 2. At least 1 episode of fecal incontinence per week. 3. History of retentive posturing or excessive volitional stool retention. 4. History of painful or hard bowel movements. 5. Presence of a large fecal mass in the rectum. 6. History of large diameter stools that may obstruct the toilet).
3. Normal Thyroid function test and negative celiac serology (IgA or IgG in patients with IgA deficiency), and no evidence of elevated RAST test for milk.
4. Parents or tutors signed informed consent to the child's participation the study.
5. Willingness to comply with the protocol.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Increase in stool number/week to at least 4 bowel movements | 8 weeks
  The measurement will be done by phone interview at week 1 and 3, and at clinic visits at week 2 and 4.
  A follow-up phone interview after the medication/placebo is stopped, at weeks 6 and 8 post enrolment.

SECONDARY OUTCOMES:
Improved stool consistency- measured by Bristol Stool Scale | 4 weeks
Improved defecation pain - measured as reduction of a pain score of 0-4 at clinic visits 2 and 4. | 4 -8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba medical center, Ramat Gan, Tel Hashomer
  - Asaf Harofe medical center, Zrifin